CLINICAL TRIAL: NCT06699030
Title: A New Strategy for Gallstone Expulsion Through Dietary Therapy: A Prospective, Single-Center, Double-Blind, Randomized Controlled Trial
Brief Title: A Strategy for Gallstone Expulsion Through Dietary Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gallstone Expulsion
Record Dates: First submitted 2024-11-16; First posted 2024-11-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Gallbladder Stone
Keywords: Gallstone; Gallbladder Function; Cholecystitis; Ultrasound Examination
MeSH Terms: conditions — Cholecystolithiasis; Gallstones; Cholecystitis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional fatty acids (Experimental): Oral Administration of functional fatty acids
  Interventions: Drug: Functional fatty acids
- Placebo (Placebo Comparator): Oral Administration of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Functional fatty acids — Days 1-3: Oral Administration of functional fatty acids Days 4-6: Oral Administration of functional fatty acids
  Arms: Functional fatty acids
Other: Placebo — Days 1-3: Placebo Days 4-6: Oral Administration of functional fatty acids
  Arms: Placebo

SUMMARY:
This study is a double-blind, prospective, single-center controlled trial conducted at a tertiary hospital, aiming to determine whether dietary therapy can effectively expel gallstones.

DETAILED DESCRIPTION:
Gallstones are a common clinical condition, and their prevalence has been increasing globally in recent years. Gallstone formation is a result of various combined factors, and in its early stages, gallstones often exist in a sludge-like form. Currently, there is no definitive research on whether gallbladder sludge can be effectively expelled through medication or dietary therapy. Therefore, the investigators are conducting a double-blind, prospective, single-center controlled trial to verify whether gallbladder sludge-like stones can be effectively expelled using dietary therapy.

ELIGIBILITY:
Inclusion Criteria:

* Gallbladder sludge-like stones with a maximum stone diameter of less than 2 mm

Exclusion Criteria:

* History of ERCP (Endoscopic Retrograde Cholangiopancreatography)
* Previous gallstone removal surgery with gallbladder preservation
* History of acute or chronic pancreatitis, cholangitis
* Mirizzi Syndrome
* History of gastrointestinal surgery
* Gastrointestinal obstruction
* Dysfunction of the sphincter of Oddi
* Gallbladder neck polyps
* Abnormal gallbladder structure
* Gallbladder mass
* Biliary infection or stones
* Congenital biliary abnormalities
* Biliary injury or surgery
* Biliary tumors
* Gastrointestinal bleeding, liver cirrhosis, or other malignant diseases
* Significant arrhythmia, bradycardia, or atrioventricular block
* Severe hypertension, liver or kidney insufficiency
* Immune, endocrine, hematological, or mental disorders
* Severe cerebrovascular disease
* Allergy to relevant foods
* Pregnant or breastfeeding women
* Unwillingness or inability to consent to participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete expulsion of gallbladder sludge after three days of intervention | 7 days
  Determined by ultrasound examination before and after the intervention to assess whether gallbladder sludge has been fully expelled
2）Number of patients with complete expulsion of gallbladder sludge after six days of intervention | 7 days
  Determined by ultrasound examination before and after the intervention to assess whether gallbladder sludge has been fully expelled

SECONDARY OUTCOMES:
Gallbladder Volume | 7 days
  Measured by ultrasound (L × W × D × 0.52)
Gallbladder Wall Thickness | 7 days
  Measured by ultrasound, accurate to 0.1 mm
Serum bilirubin | 7 days
  Determined by lab examination within 3.4-17.1μmol/L
Presence of Abdominal Pain Post-Intervention | 7 days
  If abdominal pain is present, it will be assessed using the Numerical Rating Scale (NRS) within 0-10, The higher the score, the more serious it is
Occurrence of Acute Pancreatitis Post-Intervention | 14 days
  Pain and Amy >3times as normal
Occurrence of Gastrointestinal Bleeding Post-Intervention | 14 days
  Black stool or decrease of HB
Nausea, Vomiting, and Diarrhea Post-Intervention | 14 days
  Frequency of Nausea, Vomiting, and Diarrhea Post-Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Long Deng, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhuang Q, Cheng J, Xia J, Ning M, Wu S, Shen S, Shi Y, Huang D, Dong Z, Wan X. Gypenosides Prevent and Dissolve Cholesterol Gallstones by Modulating the Homeostasis of Cholesterol and Bile Acids. Front Med (Lausanne). 2022 Apr 4;9:818144. doi: 10.3389/fmed.2022.818144. eCollection 2022. PMID 35445045
- [Background] Mulliri A, Menahem B, Alves A, Dupont B. Ursodeoxycholic acid for the prevention of gallstones and subsequent cholecystectomy after bariatric surgery: a meta-analysis of randomized controlled trials. J Gastroenterol. 2022 Aug;57(8):529-539. doi: 10.1007/s00535-022-01886-4. Epub 2022 Jun 15. PMID 35704084